CLINICAL TRIAL: NCT04414059
Title: Complications Risk Factors in Patients Hospitalized for COVID-19 Infection: Role of Proteins Electrophoresis
Brief Title: Protein Electrophoresis as a Tool for Complications Prediction in COVID-19 Hospitalised Patients
Acronym: COVELEC
Status: Completed | Type: Observational
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Other Study IDs: COVELEC; 2020-A01376-33 (Other: ID-RCB)
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: SARS-CoV 2; Hospitalisation-Associated Infection
Keywords: COVID-19
MeSH Terms: conditions — Cross Infection; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The inflammation is central in COVID-19 infections. Our aim is to evaluate the clinical value of measuring inflammation by using serum protein electrophoresis (SPE). SPE evaluation of inflammation should be able to predict outcome, follow up evolution or treatment efficacy in patients with coronavirus infection and thus anticipate their evolution to severe viral infection and allow an optimal clinical management. SPE inflammation diagnostics will be benchmarked with other diagnostics of inflammation, currently used more routinely.

DETAILED DESCRIPTION:
In late December 2019, an outbreak of an emerging respiratory disease (COVID-19) caused by a novel coronavirus named SARS-CoV-2 began in Wuhan City, Hubei Province, China and quickly spread in a substantial number of countries. The epidemic was declared a pandemic by the Word Health Organization (WHO) on 12 March 2020. SARS-CoV-2 has demonstrated the capability to spread rapidly, leading to significant impacts on healthcare systems and causing societal disruption.

Both clinical and epidemiological features of patients with COVID-19 have recently been reported, demonstrating that the SARS-CoV-2 infection can be asymptomatic in some cases or symptomatic in others. Symptomatology usually begins as mild with fever, fatigue, dry cough, and occasional dyspnea. In a minority of patients, a sudden onset of severe symptoms may develop 5-8 days into the illness including shortness of breath, pneumonitis, acute respiratory distress syndrome (ARDS) and multi organ dysfunction leading to intensive care unit (ICU) admission and high mortality. In some cases, accumulating evidence suggests that severe COVID-19 symptoms could be due to a cytokine storm syndrome. As of May 3rd 2020, the virus had infected 3,349,786 patients worldwide with more than 238,600 deaths, more often among older patients with underlying health conditions.

With caseloads overwhelming hospitals and resources stretched thin in this surging pandemic (high demand for oxygen, prolonged ventilation and even extracorporeal membrane oxygenation (ECMO), particularly for patients with acute ARDS), there is an urgent need to enhance clinical skills in order to predict from the many mild cases those few that will progress to critical illness allowing a more efficient resource allocation and clinical management.

Several studies on patient blood have described features that were most predictive of ARDS. These studies showed that severe cases, compared to mild cases, had : 1) older age; 2) abnormalities in chest scanning (CT) such as multiple patch-like shadows and ground glass opacity; 3) organ and coagulation dysfunction with a higher levels of alanine aminotransferase (ALT), lactate dehydrogenase (LDH), C-reactive protein (CRP), ferritin and D-dimer; 4) as well as markedly higher levels of immunological characteristics such as IL-2R, IL-6, IL-10, and TNF- α ; 5) and an absolute T lymphocytes (CD4+ and CD8+ T cells) number markedly lower in nearly all severe cases. These observations suggest that severity and mortality might be due to virally driven systemic hyperinflammation secondary to failure of the immune response to control infection (as shown for other viruses).

With this study we want to caracterize the predictive performance of the serum inflammation profiles by protein electrophoresis, associated with clinical, radiological and biological risk factors for worsening. This study is a prospective, observational study conducted on patients hospitalized for an infection with the SARS-CoV-2 virus.

ELIGIBILITY:
Inclusion Criteria:

* Male of female aged 18 or over
* Patients with at least one of the following diagnostic criteria, allowing to suspect an infection by the virus SARS-CoV- 2 :

  * Clinical picture with fever, and/or exertional dyspnea, and/or PO2 < 80mmHg
  * And/or chest scanner very suggestive or compatible with a COVID-19 infection
  * And/or a RT-PCR positive result already known
* Hospitalized patient in a COVID-19 medical unit, based on one or several diagnostic elements described
* Possibility to collect blood and urine samples as described in protocol
* Patients informed of the study, having understood it, and who didn't oppose to their participation

Exclusion Criteria:

* Clinical condition justifying immediate hospitalization in the intensive care unit
* During the initial patient management, an immediate need of oxygen requiring intubation and/or oxygen supply greater than 6 liters / minute
* Patients under legal protection
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥ 18 years old hospitalized in a Covid-19 medical unit for a suspected or confirmed SARS-CoV2 infection.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-09-10 (Actual)

PRIMARY OUTCOMES:
Complications onset | Up to 3 weeks
  hospitalisation in Intensive Care Unit OR Oxygen needs > 6 L/min OR death whatever the cause

SECONDARY OUTCOMES:
Risk value associated with each risk factor as identified at the end of the main study analysis | Up to 3 weeks
  Risk quantification
Predictive performance and risk associated with each individual protein fraction | Up to 3 weeks
  Correlation between complications onset (as defined by hospitalisation in Intensive Care Unit OR Oxygen needs > 6 L/min OR death whatever the cause) and individual protein fraction value
Intra-patient kinetics evolution of the electrophoresis curves | Up to 3 weeks
  Evolution over time of the serum quantity of each individual protein fraction (6 fractions studied)
Intra-patient kinetics evolution of biological risk factors | Up to 3 weeks
  Evolution over time of the serum quantity of each biological risk factor (as defined for the study)
Inter-expert reproducibility analysis of electrophoretic inflammatory profiles centrally reviewed | After study completion, estimated 10 months after first patient enrolled
  Central review of each serum protein electrophoresis curve
Contribution of urinary electrophoresis inflammation profiles in the interpretation of serum electrophoresis curves | Up to 3 weeks
  Urine samples at admission, every 4 days and at complications onset
Exploratory biological objective: Definition of a more detailed electrophoretic inflammatory profile | After study completion, estimated 10 months after first patient enrolled
  Biobank with serum samples for the implementation, at the end of the study, of a high-resolution capillary electrophoresis technique enabling each serum protein to be viewed individually

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Clinique de l'Estrée, Stains
  - Clinique Vauban, Valenciennes

REFERENCES:
- [Background] Lai CC, Shih TP, Ko WC, Tang HJ, Hsueh PR. Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and coronavirus disease-2019 (COVID-19): The epidemic and the challenges. Int J Antimicrob Agents. 2020 Mar;55(3):105924. doi: 10.1016/j.ijantimicag.2020.105924. Epub 2020 Feb 17. PMID 32081636
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Xu XW, Wu XX, Jiang XG, Xu KJ, Ying LJ, Ma CL, Li SB, Wang HY, Zhang S, Gao HN, Sheng JF, Cai HL, Qiu YQ, Li LJ. Clinical findings in a group of patients infected with the 2019 novel coronavirus (SARS-Cov-2) outside of Wuhan, China: retrospective case series. BMJ. 2020 Feb 19;368:m606. doi: 10.1136/bmj.m606. PMID 32075786
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Del Rio C, Malani PN. 2019 Novel Coronavirus-Important Information for Clinicians. JAMA. 2020 Mar 17;323(11):1039-1040. doi: 10.1001/jama.2020.1490. No abstract available. PMID 32022836
- [Background] Cheng Y, Luo R, Wang K, Zhang M, Wang Z, Dong L, Li J, Yao Y, Ge S, Xu G. Kidney disease is associated with in-hospital death of patients with COVID-19. Kidney Int. 2020 May;97(5):829-838. doi: 10.1016/j.kint.2020.03.005. Epub 2020 Mar 20. PMID 32247631
- [Background] Pei G, Zhang Z, Peng J, Liu L, Zhang C, Yu C, Ma Z, Huang Y, Liu W, Yao Y, Zeng R, Xu G. Renal Involvement and Early Prognosis in Patients with COVID-19 Pneumonia. J Am Soc Nephrol. 2020 Jun;31(6):1157-1165. doi: 10.1681/ASN.2020030276. Epub 2020 Apr 28. PMID 32345702
- [Background] Zhang X, Cai H, Hu J, Lian J, Gu J, Zhang S, Ye C, Lu Y, Jin C, Yu G, Jia H, Zhang Y, Sheng J, Li L, Yang Y. Epidemiological, clinical characteristics of cases of SARS-CoV-2 infection with abnormal imaging findings. Int J Infect Dis. 2020 May;94:81-87. doi: 10.1016/j.ijid.2020.03.040. Epub 2020 Mar 20. PMID 32205284
- [Background] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Background] Sun D, Li H, Lu XX, Xiao H, Ren J, Zhang FR, Liu ZS. Clinical features of severe pediatric patients with coronavirus disease 2019 in Wuhan: a single center's observational study. World J Pediatr. 2020 Jun;16(3):251-259. doi: 10.1007/s12519-020-00354-4. Epub 2020 Mar 19. PMID 32193831
- [Background] Chen G, Wu D, Guo W, Cao Y, Huang D, Wang H, Wang T, Zhang X, Chen H, Yu H, Zhang X, Zhang M, Wu S, Song J, Chen T, Han M, Li S, Luo X, Zhao J, Ning Q. Clinical and immunological features of severe and moderate coronavirus disease 2019. J Clin Invest. 2020 May 1;130(5):2620-2629. doi: 10.1172/JCI137244. PMID 32217835
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Background] Lee N, Chan MC, Lui GC, Li R, Wong RY, Yung IM, Cheung CS, Chan EC, Hui DS, Chan PK. High Viral Load and Respiratory Failure in Adults Hospitalized for Respiratory Syncytial Virus Infections. J Infect Dis. 2015 Oct 15;212(8):1237-40. doi: 10.1093/infdis/jiv248. Epub 2015 Apr 22. PMID 25904604
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] O'Connell TX, Horita TJ, Kasravi B. Understanding and interpreting serum protein electrophoresis. Am Fam Physician. 2005 Jan 1;71(1):105-12. PMID 15663032
- [Background] Szymanowicz A, Cartier B, Couaillac JP, Gibaud C, Poulin G, Riviere H, Le Carrer D; Groupe de Travail du College National de Biochimie des Hopitaux. [A proposal of ready-made interpretative comments applicable to serum protein electrophoresis]. Ann Biol Clin (Paris). 2006 Jul-Aug;64(4):367-80. French. PMID 16829482
- [Background] Concato J, Peduzzi P, Holford TR, Feinstein AR. Importance of events per independent variable in proportional hazards analysis. I. Background, goals, and general strategy. J Clin Epidemiol. 1995 Dec;48(12):1495-501. doi: 10.1016/0895-4356(95)00510-2. PMID 8543963
- [Background] Peduzzi P, Concato J, Feinstein AR, Holford TR. Importance of events per independent variable in proportional hazards regression analysis. II. Accuracy and precision of regression estimates. J Clin Epidemiol. 1995 Dec;48(12):1503-10. doi: 10.1016/0895-4356(95)00048-8. PMID 8543964
- [Background] Kim ES, Chin BS, Kang CK, Kim NJ, Kang YM, Choi JP, Oh DH, Kim JH, Koh B, Kim SE, Yun NR, Lee JH, Kim JY, Kim Y, Bang JH, Song KH, Kim HB, Chung KH, Oh MD; Korea National Committee for Clinical Management of COVID-19. Clinical Course and Outcomes of Patients with Severe Acute Respiratory Syndrome Coronavirus 2 Infection: a Preliminary Report of the First 28 Patients from the Korean Cohort Study on COVID-19. J Korean Med Sci. 2020 Apr 6;35(13):e142. doi: 10.3346/jkms.2020.35.e142. PMID 32242348
- [Background] Richardson S, Hirsch JS, Narasimhan M, Crawford JM, McGinn T, Davidson KW; the Northwell COVID-19 Research Consortium; Barnaby DP, Becker LB, Chelico JD, Cohen SL, Cookingham J, Coppa K, Diefenbach MA, Dominello AJ, Duer-Hefele J, Falzon L, Gitlin J, Hajizadeh N, Harvin TG, Hirschwerk DA, Kim EJ, Kozel ZM, Marrast LM, Mogavero JN, Osorio GA, Qiu M, Zanos TP. Presenting Characteristics, Comorbidities, and Outcomes Among 5700 Patients Hospitalized With COVID-19 in the New York City Area. JAMA. 2020 May 26;323(20):2052-2059. doi: 10.1001/jama.2020.6775. PMID 32320003
- See also: Coronavirus disease situation report from the WHO (3 May 2020) — https://www.who.int/docs/default-source/coronaviruse/situation-reports/20200503-covid-19-sitrep-104.pdf?sfvrsn=53328f46_4
- See also: Caution on kidney dysfunctions of 2019-nCoV patients. — https://www.medrxiv.org/content/10.1101/2020.02.08.20021212v2
- See also: Towards an Artificial Intelligence Framework for Data-Driven Prediction of Coronavirus Clinical Severity — http://techscience.com/cmc/v63n1/38464
- See also: Communiqué de presse de la Direction Générale de la Santé (29 Avril 2020) — https://solidarites-sante.gouv.fr/IMG/pdf/point_de_situation_coronavirus_du_29_avril.pdf
- See also: Coronavirus : la mortalité en réanimation beaucoup plus forte qu'annoncée en France (article du journal Le Monde du 27 Avril 2020) — https://www.lemonde.fr/planete/article/2020/04/27/coronavirus-la-mortalite-en-reanimation-beaucoup-plus-forte-qu-annoncee-en-france_6037853_3244.html